CLINICAL TRIAL: NCT01307163
Title: Systemic Variables in the Saliva of Children Undergoing Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: DR. Esti Davidovich, Hadassah Medical Organization
Other Study IDs: ran19-HMO-CTIL; esti19
Record Dates: First submitted 2008-01-10; First posted 2011-03-02 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2007-12

CONDITIONS: Liver Transplant
Keywords: saliva; liver transplantation; children; In this prospective study 60 subjects will be examined; children and adolescents; after a successful liver transplantation; informed consent forms signed be the examinees parents

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — saliva
Oversight: Data Monitoring Committee: No

SUMMARY:
Saliva is used nowadays as a significant diagnostic tool due to the latest technological developments. The research compares two experimental groups; children after liver transplantation and a control group.

Our objective is to identify from all the parameters that are evaluated, the ones that differ between the two groups. If such parameters will be found and differ statistically, it will be possible to create a non invasive medical examination protocol, which will probably be much more complaint, and being so would help locate individuals in risk groups with the tendency to develop an end-organ liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Children after a successful liver transplantation

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In this prospective study 60 subjects will be examined. Children and adolescents from Schnaidder's hospital for children after a successful liver transplantation will be characterized as the study group. As a control group, 32 healthy examinees in the same age group will be selected from the dental pediatric department at Hadassah hospital, Ein karem, Jerusalem
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization IRB, Jerusalem, Israel